CLINICAL TRIAL: NCT04679675
Title: Self-Testing Options in the Era of Primary HPV Screening for Cervical Cancer: the STEP Trial
Brief Title: Self-Testing Options in the Era of Primary HPV Screening for Cervical Cancer Trial
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Washington (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00002344; R01CA240375 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Uterine Cervical Neoplasm; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Uterine Cervical Diseases; Uterine Diseases; Cervical Cancer; Cervical Dysplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma; HPV Infection; HPV-Related Malignancy
Keywords: Cancer Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Uterine Cervical Diseases; Uterine Diseases; Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The investigators will test interventions separately by prior cervical cancer screening behavior: Screening Adherent, Overdue, and Unknown history. Interventions will differ by screening behavior.
  Previously Adherent: Previously screened for cervical cancer with a known due date within three months
  Overdue: Never screened for cervical cancer; or HPV and Pap co-test >5.25 years ago [or Pap alone >3.25 years ago]; or no past Pap and continuously enrolled at Kaiser Permanente Washington for ≥3.25 years.
  Unknown Prior Screening Behavior: Enrolled at Kaiser Permanente Washington for ≥6 months and <3.25 years, with no recorded cervical cancer screening history.
  Cohort randomization allocation will be assigned as follows to intervention arms: Previously Adherent (Usual Care, Education, Opt-in, and Direct Mail); Overdue (Usual Care, Education, and Direct Mail); and Unknown (Usual Care, Education, and Opt-in).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care
- Education (Active Comparator)
  Interventions: Behavioral: Education
- Direct Mail (Active Comparator)
  Interventions: Behavioral: Direct Mail
- Opt-in (Active Comparator)
  Interventions: Behavioral: Opt-in

INTERVENTIONS:
Other: Usual Care — Subjects will receive Kaiser Permanente Washington standard of care.
  Arms: Usual Care
Behavioral: Education — Participants will receive an Educational Brochure describing why screening for cervical cancer is important, information about HPV and its role in cervical cancer, and different strategies for cervical cancer screening.
  Arms: Education
Behavioral: Direct Mail — Participants will receive an Educational Brochure describing why screening for cervical cancer is important, information about HPV and its role in cervical cancer, and different strategies for cervical cancer screening. Participants will also receive an insert describing the home-based cervical cancer screening option and that a kit will be sent within 1 week. An HPV self-collection kit with instructions and a pre-paid return envelope (to Kaiser Permanente Washington's laboratory) will be sent to individuals with instructions on how to complete the kit.
  Arms: Direct Mail
Behavioral: Opt-in — Participants will receive an Educational Brochure describing why screening for cervical cancer is important, information about HPV and its role in cervical cancer, and different strategies for cervical cancer screening. Participants will receive an Opt-in Insert describing the home-based cervical cancer screening option and how to request a kit. Individuals can request a kit by phone or through a webpage. Individuals who request a kit will receive the HPV self-collection kit with instructions and a pre-paid return envelope (to Kaiser Permanente Washington's laboratory) will be sent to individuals with instructions on how to complete the kit.
  Arms: Opt-in

SUMMARY:
The Self-Testing options in the Era of Primary HPV screening for cervical cancer (STEP) trial will evaluate effectiveness of home-based HPV kits for improving cervical cancer screening uptake and its cost-effectiveness. The investigators will compare cervical cancer screening uptake within six months among women randomized to different outreach approaches based on prior screening behavior: A) Adherent and coming due: direct mail HPV kit vs. opt-in HPV kit vs. education; B) Overdue: direct mail HPV kit vs. education; C) Unknown: opt-in HPV kit vs. education.

DETAILED DESCRIPTION:
The scientific objective of the proposed research is to study whether an in-home programmatic HPV screening outreach strategy improves cervical cancer screening initiation and uptake. Identifying new, patient-centered options that motivate continued screening initiation and uptake is essential now and in the future.

In August 2018, the US Preventive Services Task Force released updated cervical cancer screening guidelines that include human papillomavirus (HPV) testing alone (ie, primary HPV screening) as a newly recommended strategy for women aged 30-65 years. With primary HPV screening, home-based screening is an emerging option, because HPV tests (unlike Pap tests) can be performed on clinician- or self-collected samples. Self-collected samples are as sensitive as clinician-collected samples in detecting HPV and mailing HPV self-sampling kits increases screening participation. As US healthcare systems prepare to implement primary HPV screening, they will need to consider a variety of strategies. To date, HPV self-sampling randomized clinical trials have included only overdue women; no study has evaluated uptake and acceptance of HPV self-sampling kits as an alternative to in-clinic screening in a screening-adherent population.

Based on our Home-based Options to Make cervical cancer screening Easy (HOME) trial (ClinicalTrials.gov, NCT02005510), most women will test negative (88%) and can continue routine screening; 11% will require in-clinic follow-up: 3% directly to colposcopy (HPV-16/18+ results) and 8% to Pap because of "HPV+ other" results or an unsatisfactory result (<1%). For home-based HPV screening strategies to be successful, ensuring high follow-up compliance in the minority of women who test positive is critical.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at Kaiser Permanente Washington
* Female sex
* 30 years to 64 years of age
* An intact cervix
* Has a primary care provider at Kaiser Permanente Washington

Exclusion Criteria:

* Anyone flagged by the delivery system as being on a non-routine screening schedule
* Previously randomized to the intervention arm of the HOME trial or invited to the PATH study (Participants from the PATH study and individuals randomized to the intervention arm in the HOME Study are excluded from STEP because their prior inclusion in a STEP-related research study could influence their screening uptake and affect the outcome of this trial.)
* On "do not contact list" for research studies
* Currently pregnant or had a pregnancy-related procedure within prior 3 months
* Language interpreter needed

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32771 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD, MPH, Principal Investigator — Kaiser Permanente; Rachel L Winer, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Resources developed during the study will be made available in accordance with the NIH Data Sharing Policy to researchers in both the private and public sector free or for a nominal charge and with minimal restriction. Deidentified data will be made available to qualified investigators within 6 months of acceptance of the manuscript describing major outcomes. Requestors will be required to obtain IRB approval and sign a data use agreement before data will be released. The data use agreement must include the following commitments: a commitment to using the data for research purposes only and not to identify any individual participants or to disclose Kaiser Permanente proprietary information; a commitment to securing the data using appropriate computer technology; a commitment to destroying or returning the data after analyses are completed; and a commitment to meet any additional requirements that might be stipulated by Kaiser Permanente's Human Subjects Review Committee.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Tiro JA, Metcalfe S, Muthukrishnan M, Jose A, Hansen K, Lin J, Dorsey CN, Gao H, Lacey C, Anderson ML, Meenan RT, Green BB, Buist DSM, Sparks A, Winer RL. Promoting cervical cancer screening via a mailed HPV self-collection kit: Reactions from screeners and non-screeners. Patient Educ Couns. 2026 Jan;142:109374. doi: 10.1016/j.pec.2025.109374. Epub 2025 Oct 3. PMID 41067140
- [Derived] Winer RL, Lin J, Anderson ML, Tiro JA, Green BB, Gao H, Meenan RT, Hansen K, Sparks A, Buist DSM. Strategies to Increase Cervical Cancer Screening With Mailed Human Papillomavirus Self-Sampling Kits: A Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1971-1981. doi: 10.1001/jama.2023.21471. PMID 38015219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Education | Direct Mail | Opt-in
Started | 12709 | 9279 | 2974 | 7809
Completed | 12142 | 8854 | 2897 | 7462
Not Completed | 567 | 425 | 77 | 347
Not completed — Excluded from analysis, recent Papanicolaou test prior to randomization date | 356 | 261 | 50 | 210
Not completed — Excluded from analysis, recent disenrollment from KPWA | 211 | 164 | 27 | 137

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Education | Direct Mail | Opt-in | Total
Number analyzed (Participants) | 12142 | 8854 | 2897 | 7462 | 31355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12142 | 8854 | 2897 | 7462 | 31355
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.3) | 45.6 (10.4) | 47.5 (10.0) | 45.1 (10.5) | 45.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12142 | 8854 | 2897 | 7462 | 31355
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 628 | 502 | 154 | 421 | 1705
  Not Hispanic or Latino | 8047 | 5278 | 2307 | 4446 | 20078
  Unknown or Not Reported | 3467 | 3074 | 436 | 2595 | 9572
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 76 | 50 | 16 | 41 | 183
  Asian | 1298 | 919 | 326 | 861 | 3404
  Native Hawaiian or Other Pacific Islander | 153 | 120 | 30 | 69 | 372
  Black or African American | 553 | 411 | 133 | 315 | 1412
  White | 7175 | 4844 | 1902 | 4176 | 18097
  More than one race | 353 | 261 | 92 | 208 | 914
  Unknown or Not Reported | 2534 | 2249 | 398 | 1792 | 6973
Region of Enrollment [Number; unit: participants]
  United States | 12142 | 8854 | 2897 | 7462 | 31355

OUTCOME MEASURES:

1. Primary Outcome: Screening Completion by Outreach Approach and Prior Screening Behavior
Description: Rate of completing cervical cancer screening completion by outreach approach and prior screening behavior. Screening completion defined by returning the home kit and attending the recommended in clinic follow-up (if applicable); or receiving in clinic screening.
Time Frame: Within 6 months of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Education | Direct Mail | Opt-in
Number analyzed (Participants) | 12142 | 8854 | 2897 | 7462
Participants
  Screening-Adherent | 3671 | 3960 | 1482 | 3956
  Overdue | 5488 | 1408 | 1415 | 0
  Unknown | 2983 | 3486 | 0 | 3506
Statistical Analysis 1: Comparison: Education vs Direct Mail; Primary analysis stratified by screening history. These results are for Screening-Adherent (population):Direct-Mail versus Education analysis; Test type: Superiority; p = 0.05, Poisson Regression with GEE; Risk Ratio (RR) = 1.30, 95% CI 2-sided [1.23 to 1.36]
Statistical Analysis 2: Comparison: Education vs Opt-in; Primary analysis stratified by screening history. These results are for Screening-Adherent (population):Opt-In versus Education analysis; Test type: Superiority; p = .05, Poisson Regression with GEE; Risk Ratio (RR) = 1.07, 95% CI 2-sided [1.02 to 1.12]
Statistical Analysis 3: Comparison: Education vs Direct Mail; Primary analysis stratified by screening history. These results are for Screening-Overdue (population):Direct-Mail versus Education analysis; Test type: Superiority; p = .05, Poisson Regression with GEE; Risk Ratio (RR) = 1.90, 95% CI 2-sided [1.68 to 2.16]
Statistical Analysis 4: Comparison: Education vs Opt-in; Primary analysis stratified by screening history. These results are for Screening-Unknown (population):Opt-In versus Education analysis; Test type: Superiority; p = .05, Poisson Regression with GEE; Risk Ratio (RR) = 1.14, 95% CI 2-sided [1.03 to 1.25]

2. Secondary Outcome: Incremental Cost-effectiveness Ratio by Outreach Approach and Prior Screening Behavior
Description: Incremental cost-effectiveness ratio, which will be defined for each outreach approach within each screening behavior subgroup. Also, comparisons across screening behavior subgroups of usual care plus education to usual care.
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

3. Secondary Outcome: Screening Initiation by Outreach Approach and Prior Screening Behavior
Description: Screening Initiation defined as returning the home kit or receiving in clinic cervical cancer screening.
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

4. Secondary Outcome: Time From Randomization to Screening Completion by Outreach Approach and Prior Screening Behavior
Description: Time from randomization to screening completion by outreach approach and prior screening behavior. Screening completion defined by returning the home kit and attending the recommended in clinic follow-up (if applicable); or receiving in clinic screening.
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

5. Secondary Outcome: Completion of Recommended Follow-up After a Positive Kit Result
Description: Proportion of intervention group women who complete recommended follow-up after a positive kit result by outreach approach and prior screening behavior. Per current guidelines, in-clinic Pap after other-HR HPV positive; or colposcopy after HPV 16/18+ HPV self-collection
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

6. Secondary Outcome: Screening Method Choice
Description: Proportion of intervention group women who do not screen, return the home kit or receive in-clinic screening by outreach approach and prior screening behavior. Screening uptake outcome (no screen, home kit, or in-clinic) by outreach approach and by prior screening behavior
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

7. Secondary Outcome: Qualitative Information From Focus Groups on Patient Preferences by Prior Screening Behavior
Description: Through focus groups, the investigators will explore patient preference for, and satisfaction with, home HPV screening and barriers to follow-up of abnormal screening results.
Time Frame: 6-12 months following study invitation
Reporting Status: Not Posted

8. Secondary Outcome: Health System Costs to Implementing Home Testing by Outreach Approach and Prior Screening Behavior
Description: Economic assessment of system-level financial consequences of adopting home-based HPV screening for cervical cancer. These analyses will evaluate the needed time to follow-up for the next cervical cancer screening to reduce gaps in cervical cancer screening HEDIS metrics, which also addresses program affordability.
Time Frame: 3-5 years (projected)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected within 6 months of randomization.
Description: Usual Care and Education arm participants are not at risk for adverse events because they did not use, nor have the option to use, a self-collect screening kit.
Arm/Group | Usual Care | Education | Direct Mail | Opt-in
All-Cause Mortality (participants affected / at risk) | 0/12142 | 0/8854 | 0/2897 | 0/7462
Serious Adverse Events (participants affected / at risk) | 0/12142 | 0/8854 | 0/2897 | 0/7462
Other Adverse Events (participants affected / at risk) | 0/12142 | 0/8854 | 4/2897 | 3/7462
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=12142) | Education (N=8854) | Direct Mail (N=2897) | Opt-in (N=7462)
Dysuria (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04679675/Prot_SAP_000.pdf